CLINICAL TRIAL: NCT00185146
Title: Effect of Pactimibe on the Progression of Atherosclerosis as Measured by 2-D and 3-D Carotid Ultrasound
Brief Title: Efficacy and Safety of Pactimibe in Patients With Atherosclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sankyo Pharma Gmbh (Industry)
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SE-505/14
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-03-28 (Estimated); Status verified 2007-03

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — pactimibe

INTERVENTIONS:
Drug: Pactimibe

SUMMARY:
The effect of pactimibe on the reduction of atherosclerosis in the carotid artery will be assessed using carotid ultrasound

ELIGIBILITY:
Inclusion Criteria:

* Increased cardiovascular risk (i.e. history of myocardial infarction, stroke, diabetes mellitus, left ventricular hypertrophy)
* Intima-media thickness greater than or equal to 0.8 mm as measured by ultrasonography
* Negative pregnancy test for females

Exclusion Criteria:

* Whole blood donation (greater than or equal to 450 ml) during the last three months before study start
* Unstable angina, congestive heart failure or uncontrolled hypertension
* Renal disease including nephrectomy and/or renal transplant
* Hepatic disease or abnormal liver function parameters
* Drug abuse or alcohol addiction

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-09; Study Completion 2005-08

PRIMARY OUTCOMES:
Efficacy of pactimibe versus placebo on the progression of atherosclerosis

SECONDARY OUTCOMES:
Safety and tolerability of pactimibe versus placebo in patients with atherosclerosis

CONTACTS AND LOCATIONS:
Overall Officials: P U Witte, MD, PhD, FFPM, Principal Investigator — IMFORM GmbH
Locations (1):
- Munich, Germany